CLINICAL TRIAL: NCT02671396
Title: Effects of Virtual Reality Based Training on Posture Stability in Individuals With Parkinson's Disease
Brief Title: Effects of Virtual Reality Based Training on Posture Stability in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13MMHIS120
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: Virtual Reality; Postural Stability; Balance Training; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual reality based intervention (Experimental): Virtual reality based balance training
  Interventions: Behavioral: Virtual reality based intervention
- Conventional intervention (Active Comparator): Conventional balance training
  Interventions: Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: Virtual reality based intervention — Virtual reality based balance training
  Arms: Virtual reality based intervention
Behavioral: Conventional intervention — Conventional balance training
  Arms: Conventional intervention

SUMMARY:
The present study is to examine the effects of a virtual reality based balance training using the Kinect sensor on postural stability and functional balance in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr stages I through III
* A score of more than or equal to 24 on the mini-mental state examination
* Stable medication usage
* Freedom from any other problems that might affect training

Exclusion Criteria:

* Unstable medical conditions
* Histories of other diseases known to interfere with participation in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Limits of stability test | Change from Baseline at 8 weeks
One-leg stance test | Change from Baseline at 8 weeks

SECONDARY OUTCOMES:
Berg Balance Scale | Change from Baseline at 8 weeks
Timed up and go test | Change from Baseline at 8 weeks

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shih MC, Wang RY, Cheng SJ, Yang YR. Effects of a balance-based exergaming intervention using the Kinect sensor on posture stability in individuals with Parkinson's disease: a single-blinded randomized controlled trial. J Neuroeng Rehabil. 2016 Aug 27;13(1):78. doi: 10.1186/s12984-016-0185-y. PMID 27568011